CLINICAL TRIAL: NCT07293936
Title: Validation of a Post-Filter Hematocrit Calculation Formula: A Comparative Analysis With Measured Post-Filter Hematocrit Values
Brief Title: Post-Filter Hematocrit
Acronym: CRRTHCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gwyndolyn M. Radford (Other)
Responsible Party: Sponsor-Investigator, Gwyndolyn M. Radford, Principal Investigator, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 202412294
Record Dates: First submitted 2025-03-04; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Continuous Renal Replacement Therapy; Renal Failure; Hemofilter Clotting
Keywords: crrt; continuous renal replacement therapy; hemofilter clotting; post-filter hematocrit; filtration fraction
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Intervention Model Description: All participants will undergo the same "intervention" of both using their blood samples to measure post-filter hematocrit and using their other lab values and CRRT settings to calculate post-filter hematocrit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CRRT patients (Other): All participants will receive the same "intervention" of both measuring and calculating post-filter hematocrit.
  Interventions: Other: Calculated Post-Filter Hematocrit; Other: Measured Post-Filter Hematocrit

INTERVENTIONS:
Other: Calculated Post-Filter Hematocrit — using the formula: HCTpost=HCTpre/(FF(HCTpre-1)+1)
Other: Measured Post-Filter Hematocrit — Measured from blood sample taken from CRRT machine

SUMMARY:
Filter clotting is a major complication of continuous renal replacement therapy (CRRT), resulting in blood loss, reduced treatment efficacy, and increased cost. One modifiable factor associated with filter clotting is filtration fraction (FF), or the proportion of plasma water being removed from the blood over the course of the filter. In convention, a cutoff of FF<20-30% has been used to prevent hemofilter clotting, but no evidence correlating FF with hemofilter clotting has been documented. Some experts have proposed that post-filter hematocrit (Hct) could be a more direct marker for determining hemofilter clotting risk, but evidence supporting clinical utility of this marker is lacking.

HCTpost=HCTpre/(FF(HCTpre-1)+1)

In our proposed validation study, we hope to determine whether our formula for post-filter Hct provides accurate results when compared to measured values. The information obtained from this study will potentially justify the use of utilizing the formula in future studies.

The procedure of this study is collecting blood samples from the post-filter lines of patients on CRRT at different time points and different flow rates. This will be considered the "measured post-filter hematocrit" which will then be compared to the calculated formula above, using the other values obtained from daily labs (for pre-filter hematocrit) and CRRT machine settings.

DETAILED DESCRIPTION:
This investigational study is listed as "other" because it is a validation study comparing two measurement methods-comparing a calculated versus a machine-measured post-filter hematocrit- and is typically classified as a cross-sectional investigational study in the context of diagnostic or method comparison research.

ELIGIBILITY:
Inclusion Criteria:

* patients initiated on CRRT age equal than or greater to 18 years of age

Exclusion Criteria:

* patients on ECMO

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03-15 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Agreement between measured and calculated post-filter hematocrit values. | Participation begins at consent and includes a single study procedure in which four post-filter blood samples are collected over ~40 minutes. Participation ends after the final draw. Generally, no longer than 1 day.
  Use Bland-Altman analysis to assess agreement and quantify bias and limits of agreement. Calculate correlation coefficients (Pearson or Spearman) to evaluate the strength of association.

SECONDARY OUTCOMES:
Analyze the impact of CRRT settings on discrepancies between measured and calculated Filtration Fraction | Participation begins at consent and includes a single study procedure in which four post-filter blood samples are collected over ~40 minutes. Participation ends after the final draw. Generally, no longer than one day.
  How do different settings (e.g., Q_B, Q_UF, Q_prefilter, Q_postfilter) on the machine affect the discrepancies (if there are any) between calculated and measured filtration fraction. Will be using change in post-filter hematocrit values as the measured filtration fraction and comparing to calculated filtration fraction using standard flow-rate derived formula used in practice.
Subgroup analysis based on patient-specific factors | Participation begins at consent and includes a single study procedure in which four post-filter blood samples are collected over ~40 minutes. Participation ends after the final draw.
  Post-filter hematocrit values will be stratified and compared across subgroups defined by baseline pre-filter hematocrit category, anticoagulation strategy (e.g., citrate vs. heparin vs. none), and blood-flow rate category. The metric reported will be the mean post-filter hematocrit within each subgroup and the between-group differences.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No